CLINICAL TRIAL: NCT00205257
Title: Prediction of Acute Graft Rejection by Examining Urine Chemokines in Patients With Kidney Transplant
Brief Title: Prediction of Acute Rejection in Renal Transplant
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2001-252
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2013-12

CONDITIONS: Kidney Transplant

SUMMARY:
Acute rejection is still a major risk factor affecting the prognosis of kidney transplant patients. Alloreactive cells of the recipient infiltrate the kidney graft and cause inflammatory reaction which damages the graft structure and function. Conventional diagnosis of acute rejection is based on clinical symptoms and kidney biopsy examination. The clinical symptoms are a result of the kidney damage, which occurs days after the initiation of the rejection reaction. Kidney biopsy is an invasive and expensive procedure. It has been wished to have new parameters that can replace/supplement the conventional procedures. Chemokines are small molecules that attract inflammatory cells. Changes of chemokine levels in the urine may correlate with the immune status in the kidney. A systematic study to evaluate the chemokine levels in urine and correlation with the kidney biopsy pathology will answer the question whether monitoring of urinary chemokines would be useful in predicting graft rejection/damage.

ELIGIBILITY:
Inclusion Criteria:

* One hundred subjects undergoing kidney biopsy for suspected rejection
* Forty subjects that have stable graft function with normal level of blood creatinine (No biopsy is needed at the time of sample collection).

Exclusion Criteria:

* Subjects under the age of 18
* Gender of potential subjects male or female
* Age Limits greater than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-09; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
kidney biopsy pathology | 1 year

SECONDARY OUTCOMES:
urinary chemokines | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Chin, Principal Investigator — University of Wisconsin Medical School